CLINICAL TRIAL: NCT01140113
Title: Does Modified Ultrafiltration Improves Inflammatory Response and Cardiopulmonary Function After CABG Procedures?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Campinas, Brazil (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Orlando Petrucci, MD, PhD, University of Campinas, Brazil
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Modified Ultrafiltration
Record Dates: First submitted 2010-06-07; First posted 2010-06-09 (Estimated); Last update posted 2013-07-23 (Estimated); Status verified 2013-07

CONDITIONS: Coronary Artery Disease; Cardiac Surgical Procedures
Keywords: hemoconcentration; ultrafiltration; coronary artery disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Ultrafiltration

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (No Intervention): this group had undergone to routine coronary artery bypass graft surgery
- Modified Ultrafiltration (Experimental): patients after weaning from bypass were submitted to ultrafiltration
  Interventions: Procedure: Modified Ultrafiltration

INTERVENTIONS:
Procedure: Modified Ultrafiltration — After weaning from bypass patients had undergone to modified ultrafiltration for 15 minutes with a filtration flow at 300 ml/min
  Other Names: Ultrafiltration
  Arms: Modified Ultrafiltration

SUMMARY:
The inflammatory response after cardiac surgery increases mortality and morbidity. Modified ultrafiltration (MUF) has been shown to decrease the post-cardiac surgery inflammatory response, to improve respiratory function, and cardiac performance in pediatric patients; however, this approach has not been well established in adults. The investigators therefore hypothesized that MUF can decrease the post-cardiac surgery inflammatory response and can improve cardiopulmonary function in adults.

DETAILED DESCRIPTION:
Patient selection After Institutional Review Board approval, a prospective study was carried out with 60 consecutive patients underwent CABG cardiopulmonary bypass (CPB) in our institution. All patients signed a consent form before enrolled into the study. The patients were randomly assigned to a control group treated with no modified ultrafiltration (CO group) or to a treatment group with modified ultrafiltration (MUF group) after bypass period. The inclusion criteria were: patients aged from 30 to 70 years old, both genders, left ventricle ejection fraction higher than 39%, normal renal function, with or without diabetes, and who underwent CABG with no associate procedures. The exclusion criteria were: left ventricle ejection fraction lower than 39% and abnormal renal function (serum creatinine > 2.0 mg/dl, clearance lower than 45 mL/m in males or lower than 40 mL/m in females).

Surgical procedure:

After anesthesia induction, the patients were monitored using a continuous cardiac output catheter (Edwards Lifesciense, Irvine. USA), invasive arterial mean pressure catheter, and urine output catheter.

All patients were submitted to tepid bypass (32 o C) with a target flow of 2.4 L/min/m2. After CPB was established the aorta was cross clamped and the distal anastomoses were performed. The blood tepid cardioplegia were used during the cross clamp period. The clamp was released and a C-clamp was applied for the proximal anastomosis effectuation. After a proximal anastomosis complementation, the patients were weaned from the bypass. Following the CPB period the patients were randomly assigned to MUF group or CO group. All operations were performed by one surgeon (O.P.).

Modified Ultrafiltration. The ultrafiltration was performed in heparinized patients between the arterial and the venous tubings of the CPB circuit, using a H-500 filter (polyestersuphone) with an effective membrane area of 0.5 m2, pore size of 5 nm, prime volume of 34 ml, maximum transmembrane pressure of 400 mmHg, internal fiber diameter of 200 µm, and fiber thickness wall of 30 µm (Braile Biomedica, São José do Rio Preto, Brazil).

The blood flow through the filter was 300 ml/min, which as maintained by a roller pump on the inlet part of the filter. Suction was applied to the filtrate port to achieve a negative pressure of 100 mmHg. The process was carried out for 15 minutes in all patients who underwent MUF while the patients assigned to CO group were observed for 15 minutes.

The hemostasis was reviewed, a mediastinal drain was inserted, the patient was closed, and sent to the intensive care unit.

Blood sample, oxygen transport, and hemodynamic parameters regimen:

The hemodynamic and oxygen transport parameters such as cardiac output index, systemic vascular resistance index, pulmonary vascular resistance index, arterial mean pressure, oxygen delivery (DO2), oxygen consumption (VO2), oxygen index (OI), and alveolar-arterial gradient (A-aDO2) were recorded.

The oxygen index was calculated by the following equation: OI = (FiO2 X MAP)/PaO2. The A-aDO2 were calculated by the equation: A-aDO2 = 713 X FiO2 - PaO2 - PaCO2). Where FiO2 is inspired fraction of oxygen, MAP is mean airway pressure, PaO2 is partial pressure of oxygen in the arterial blood, and PaCO2 is partial pressure of carbon dioxide in the arterial blood.

Blood samples were collected from arterial line with heparin coated tubes for interleukin 6 (IL-6), P-selectin, E-selectin, and intercellular adhesion molecule (ICAM) determination at the following times: after induction of anesthesia, pre MUF after bypass, post MUF, 24 hours after surgery, and 48 hours after of surgery. Blood samples were centrifuged for 20 minutes at 4oC and the serum was aliquoted and stored at - 70oC. The inflammatory markers were measured using commercially available ELISA kits (R&D Systems, Abingdon, UK).

Clinical variables:

Patients demographic data and medical history were collected prospectively. Postoperative data such as ICU length of stay (days), hospital length of stay (days), total blood loss in 48 hours, units of red blood cell transfusions, serum creatinine, international normalized ratio for prothrombin time (INR), partial thromboplastin time ratio (PR), leukocytes count, serum lactate, and urea nitrogen (BUN) were also recorded.

Statistical analyzes The continuous variables were expressed as mean with one standard deviation, the categorical variables were expressed as frequency. All data were tested for normality and the necessary transformations were performed as necessary. The t test for unpaired samples was used for total bleeding and requirements of RBC units transfusion analysis. The two-way ANOVA was performed for intragroup, intergroup, and time/group interactions with Bonferroni post-hoc test (GraphPad Prism version 5.0 for Mac OS X. San Diego California. USA). The P-values < 0.05 were considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* elective patients to coronary artery bypass graft surgery
* left ventricle ejection fraction higher than 40%

Exclusion Criteria:

* renal impairment (serum creatinine higher than 1.7 mg%)
* neoplasm

Ages: 30 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2007-07; Primary Completion 2008-07 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Overall clinical improvement after cardiac surgeries. | 30 day after surgery

SECONDARY OUTCOMES:
The treatment group has less inflammatory markers | 30 days
The treatment group has improvements in the respiratory variables | 30

CONTACTS AND LOCATIONS:
Overall Officials: Orlando Petrucci, MD, PhD, Principal Investigator — University of Campinas
Locations (1):
- Hospital da Clinicas, Campinas, São Paulo, Brazil

REFERENCES:
- [Derived] Torina AG, Silveira-Filho LM, Vilarinho KA, Eghtesady P, Oliveira PP, Sposito AC, Petrucci O. Use of modified ultrafiltration in adults undergoing coronary artery bypass grafting is associated with inflammatory modulation and less postoperative blood loss: a randomized and controlled study. J Thorac Cardiovasc Surg. 2012 Sep;144(3):663-70. doi: 10.1016/j.jtcvs.2012.04.012. Epub 2012 May 9. PMID 22578899